CLINICAL TRIAL: NCT05017831
Title: Shifting Perspectives R33 Phase: Enhancing Outcomes in Adolescent Anorexia Nervosa With Cognitive Remediation Therapy (CRT)
Brief Title: Shifting Perspectives R33 Phase: Enhancing Outcomes in Anorexia Nervosa With CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 21-019079; 5R61MH119262-02 (NIH); R33MH119262 (NIH)
Record Dates: First submitted 2021-08-03; First posted 2021-08-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Random assignment to one of two groups.
Who Masked: Outcomes Assessor
Masking Description: Any study team member who is assessing for outcomes will not know which participant/family is in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Based Treatment (FBT) (Active Comparator): Families will receive 15 sessions of FBT alone.
  Interventions: Behavioral: Family Based Treatment
- FBT w/ Adolescent-focused Cognitive Remediation Therapy (Experimental): Family Based Treatment with Adolescent-focused Cognitive Remediation Therapy (CRT): Families will receive 15 sessions of FBT over six months. The first 9 sessions of FBT will be preceded by adolescent-focused CRT.
  Interventions: Behavioral: Family Based Treatment; Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Family Based Treatment — Family Based Treatment (FBT) is an evidence based treatment in which parents are responsible for adolescent re-nourishment. They play an active role in treatment and their self-efficacy to make decisions regarding their child's treatment is empowered.
  Other Names: FBT
Behavioral: Cognitive Remediation Therapy — Cognitive Remediation Therapy (CRT) is an adjunctive treatment focused on increasing set-shifting ability and developing meta-cognition. CRT is a behavioral treatment that presents tasks to participants in a standardized order within each session. Each task has a number of levels. Participants stay at the same task-based level until mastered. They then move up a level on that task. participants can be at different levels on different tasks within each session. After completion of tasks, participants are asked to reflect on their thought processes in solving the tasks. Standard prompts are used to guide the discussion.
  Other Names: CRT
  Arms: FBT w/ Adolescent-focused Cognitive Remediation Therapy

SUMMARY:
Anorexia Nervosa is a serious life-threatening illness with a typical age of onset in adolescence; if not effectively treated, it has the potential to significantly impact adolescent development and quality of life. Research on executive functioning in anorexia nervosa indicates that it may be a viable target for intervention that could improve outcome. The current project focuses on determining whether or not the investigators can improve set-shifting in affected adolescents in the hopes that improvements in set-shifting will, ultimately, improve outcome.

DETAILED DESCRIPTION:
This is the second phase (R33) of a two-phased project exploring the effect of adding Cognitive Remediation Therapy (CRT) to traditional Family Based Treatment (FBT) for adolescents with Anorexia Nervosa (AN) and their families. This phase (R33) follows a prior 2-year study (R61) which examined the impact of CRT on set-shifting abilities (a type of executive functioning often referred to as cognitive flexibility). This second phase aims to replicate findings from the first study as well as examine whether the addition of CRT to traditional FBT will impact treatment outcomes (e.g., eating disorder symptoms, weight outcomes). CRT is an adjunctive treatment approach where adolescents learn different ways of thinking and problem solving to become more flexible thinkers. The investigators will recruit and randomly assign 96 families of youth with AN to either an FBT group or FBT with adolescent-focused CRT group. Parents and adolescents will complete questionnaires and assessments to evaluate outcomes and predictors of outcome. Evidence supporting FBT+CRT to increase set-shifting in adolescents will inform future efforts to leverage understanding of neurobiology of AN in adolescents to improve outcome. Results will also inform how best to augment current treatments, support parents, and increase positive outcomes for adolescents with AN, and reduce relapse.

ELIGIBILITY:
Inclusion Criteria: Adolescents

1. Age 12-18
2. Currently meets Diagnostic and Statistical Manual-5 criteria for Anorexia Nervosa
3. Medically stable for outpatient treatment
4. Fluent in English
5. No co-morbid condition that would exclude participation
6. Medical clearance from primary care physician and permission to speak to Primary Care Physician about clinical issues
7. Biological parent or primary caregiver willing to engage in treatment and who lives with the adolescent

Inclusion Criteria: Parents

1. Age >18
2. Child with a diagnoses of AN
3. Parent or caregiver willing to participate
4. Fluent in English
5. No co-morbid condition that would exclude participation

Exclusion Criteria: Adolescents

1. Adolescent outside age range
2. No more than four sessions of prior CRT in any format
3. Pregnant adolescent
4. Presence of: pervasive developmental disability, psychosis, bipolar disorder, substance abuse, autism spectrum disorder, or intellectual disability
5. Presence of: a brain disorder or injury (such as TBI) that could impact the ability to engage in treatment
6. Use of anti-psychotic medication during first 15 FBT sessions. Use of this medication is permitted in the optional 12 FBT sessions in the 6-month follow-up period of this study. This medication can affect cognitive abilities, which may interact with assessments that measure cognitive flexibility. However, we do not measure cognitive flexibility in the 6-month follow-up period when the 12 additional FBT sessions can take place.
7. Concurrent psychosocial therapy

Exclusion Criteria: Parents

1. Presence of: pervasive developmental disability, psychosis, uncontrolled bipolar disorder, substance abuse, autism spectrum disorder, or intellectual disability.
2. Presence of: a brain disorder or injury (such as TBI) that could impact the ability to engage in treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Change in executive functioning | Baseline, during treatment, end of treatment
  Investigators will use the Delis Kaplan Executive Functioning System (D-KEFS ) Trails Number-Letter Sequencing subtest, a neurocognitive behavioral task, to assess ability to set-shift (a core component of executive functioning). Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better executive functioning.
Change in response inhibition | Baseline, during treatment, end of treatment
  Investigators will use the Delis Kaplan Executive Functioning System Inhibition subtest, neurocognitive behavioral task, to assess ability to inhibit automatic responses. Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better response inhibition.
Change in set-shifting | Baseline, during treatment, end of treatment
  Also using the Delis Kaplan Executive Functioning System Inhibition task, investigators will use scores from the D-KEFS Inhibition/Switching subtest to assess ability to switch between alternating rules (a component of set shifting). Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better set-shifting.
Change in shifting accuracy | Baseline, during treatment, end of treatment
  Investigators will use the Delis Kaplan Executive Functioning System Verbal Fluency subtest, neurocognitive behavioral task, to assess accuracy in shifting categories (a component of executive functioning). Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better shifting accuracy.
Change in category switching flexibility | Baseline, during treatment, end of treatment
  Investigators will also use the Delis Kaplan Executive Functioning System Verbal Fluency subtest, category switching scores, to assess flexible switching (a component of executive functioning). Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better switching flexibility.
Change in flexibility | Baseline, during treatment, end of treatment
  Investigators will use the Delis Kaplan Executive Functioning System Sorting subtest, neurocognitive behavioral task, to assess changes in flexibility.Investigators will compare change in scaled scores from pre, during, and post-treatment across groups. Scaled scores range from 0-19 with higher scores indicating better flexibility.
Change in self-reported inhibition control | Baseline, during treatment, end of treatment
  The Behavior Rating Inventory of Executive Functioning is a self and parent-report measure of executive functioning. The measure comprises 10 clinical scales, of which investigators will use the Inhibition subscale to assess self-reported inhibition control (ranged from 0-100, with higher reporting greater set-shifting ability). Investigators will compare change in T scores from pre, during, and post-treatment across groups.
Change in self-reported set-shifting | Baseline, during treatment, end of treatment
  The Behavior Rating Inventory of Executive Functioning is a self and parent-report measure of executive functioning. The measure comprises 10 clinical scales, of which investigators will use the Shifting subscale to assess self-reported set-shifting. Investigators will compare change in T scores (ranged from 0-100, with higher reporting greater set-shifting ability) from pre, during, and post-treatment across groups.
Rate of weight gain | Baseline, during treatment, end of treatment
  Investigators will weigh participants during treatment to compare rate of change (slope) in weight gain from pre, during, and post-treatment across groups. Larger change in weight indicates greater recovery from the eating disorder.
Change in eating disorder symptomology | Baseline, during treatment, end of treatment
  Adolescents will complete the Eating Disorder Examination - Questionnaire (a 28-item self-report measure of eating disorders symptomatology), while parents will complete the Anorectic Behavior Observation Scale (a 30-item collateral report measure of eating and exercise behavior). Investigators will examine changes in these scores from baseline, during, and post-treatment. Scores range from 0-6 with higher scores suggesting more severe eating disorder symptomatology.
Change in behavioral flexibility (amount consumed) | Baseline, during treatment, end of treatment
  Adolescents will complete a buffet meal during which investigators will record the amount of food they consume in grams. This task aims to assess changes in behavioral flexibility by objectively assessing food choice in individuals with an eating disorder. Investigators will examine changes from baseline, during, and at treatment completion. A larger amount of food eaten (in grams) represents greater behavioral flexibility.
Change in behavioral flexibility (eating disorder behaviors) | Baseline, during treatment, end of treatment
  Adolescents will complete a buffet meal during which investigators will record eating behaviors using a novel checklist (a total score of eating disorder behaviors observed). These behaviors include staring, fidgeting, inappropriate napkin use, frequency of food tearing, frequency of dissecting food. Minimum score for this variable is 0, however, there is no maximum frequency. This task aims to assess changes in behavioral flexibility by objectively assessing eating-related behaviors in individuals with an eating disorder, with higher scores suggesting lower behavioral flexibility. Investigators will examine changes from baseline, during, and at treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Alix Timko, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timko CA, Bhattacharya A, Fitzpatrick KK, Howe H, Rodriguez D, Mears C, Heckert K, Ubel PA, Ehrenreich-May J, Peebles R. The shifting perspectives study protocol: Cognitive remediation therapy as an adjunctive treatment to family based treatment for adolescents with anorexia nervosa. Contemp Clin Trials. 2021 Apr;103:106313. doi: 10.1016/j.cct.2021.106313. Epub 2021 Feb 1. PMID 33539993
- [Background] Orloff NC, McGinley K, Lenz K, Mack AS, Timko CA. Adaptations of cognitive remediation therapy for adolescents with anorexia nervosa for delivery via telehealth. Int J Eat Disord. 2023 Jan;56(1):72-79. doi: 10.1002/eat.23850. Epub 2022 Nov 19. PMID 36401578
- [Background] Cooper M, Mears C, Heckert K, Orloff N, Peebles R, Timko CA. The buffet challenge: a behavioral assessment of eating behavior in adolescents with an eating disorder. J Eat Disord. 2024 Jan 18;12(1):8. doi: 10.1186/s40337-024-00968-3. PMID 38238787
- [Background] Miller ML, Timko CA, Hormes JM. Factor structure of the Eating Disorder Flexibility Index in U.S. nonclinical collegiate and clinical adolescent samples. Eat Behav. 2024 Jan;52:101847. doi: 10.1016/j.eatbeh.2024.101847. Epub 2024 Jan 27. PMID 38301405
- [Background] Timko CA, Schnabel J, Orloff NC. The importance of improving cognitive flexibility in adolescents with anorexia nervosa: The case for cognitive remediation therapy. Int J Eat Disord. 2024 May;57(5):1109-1118. doi: 10.1002/eat.24164. Epub 2024 Feb 9. PMID 38333943